CLINICAL TRIAL: NCT00770614
Title: Hydration and Contrast-Induced Nephropathy in Primary Angioplasty. A Randomized, Placebo Controlled, Trial.
Brief Title: Hydration and Contrast-Induced Nephropathy in Primary Angioplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Misericordia e Dolce (Other)
Responsible Party: Principal Investigator, Mauro Maioli, MD, Ospedale Misericordia e Dolce
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prato0703; POCARD0703
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast Induced Nephropathy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Sodium Bicarbonate (154 mEq/L in dextrose and H2O) 3 mL/kg for 1 hour before contrast medium, followed by an infusion of 1 mL/kg/h for 12 hours after the procedure
  Interventions: Drug: sodium bicarbonate solution
- 2 (Active Comparator): Isotonic Saline (0.9% sodium chloride) 1 mL/kg/h for 12 hours after the procedure
  Interventions: Drug: Isotonic saline
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sodium bicarbonate solution — 154 mEq/L in dextrose and H2O
  Arms: 1
Drug: Isotonic saline — 0.9% sodium chloride
  Arms: 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether hydration with sodium bicarbonate is more effective than hydration with sodium chloride to prevent contrast induced nephropathy in patients undergoing Primary Coronary Intervention for Acute ST Elevation Myocardial Infarction.

ELIGIBILITY:
Inclusion Criteria:

* patients with Acute ST Elevation Myocardial Infarction submitted to Primary Intervention

Exclusion Criteria:

* refusal to consent
* previous contrast exposure within 72 hours

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2004-03; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Absolute increase of at least 0.5 mg/dl from the baseline value in serum creatinine concentration or a relative increase ≥ 25% over baseline serum creatinine within 5 days after contrast agent administration | within 5 days after contrast exposure

SECONDARY OUTCOMES:
Adverse clinical events within 1 month, including in-hospital death and need for dialysis or hemofiltration | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maioli, MD, Principal Investigator — Ospedale Misericordia e Dolce, Prato
Locations (1):
- Ospedale Misericordia e Dolce, Prato, Prato, Italy